CLINICAL TRIAL: NCT03499015
Title: Balloon Dilation of the Eustachian Tube in Children: a Randomized Side-controlled Clinical Trial
Brief Title: Balloon Dilation of the Eustachian Tube in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Arnoldner, Assoc. Prof. PD M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK Nr: 1795/2017
Record Dates: First submitted 2018-03-25; First posted 2018-04-17 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Glue Ear; Tube Disorders Eustachian
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Intervention Model Description: single-sided treatment, contralateral side with same pathology works as control
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only surgeon knows treated side, documentation of side only visible to surgeon and investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear without BET (No Intervention): ear without BET treatment works as control
- BET ear (Experimental): ear with BET treatment works as intervention arm
  Interventions: Procedure: Balloon Eustachian Tuboplasty (BET)

INTERVENTIONS:
Procedure: Balloon Eustachian Tuboplasty (BET) — A balloon catheter is used to dilate the cartilage part of the eustachian tube and is inserted through the nose to reach the opening of the tube, located in the nasopharynx.
  Arms: BET ear

SUMMARY:
Otitis media with effusion (OME) is very common in children and characterized by fluid in the middle ear without signs or symptoms of acute ear infection. Treatment options are tympanostomy tubes and/or adenoidectomy. However OME often reoccurs after these procedures.

Goal of this study will be to evaluate the Balloon Eustachian Tuboplasty (BET) in children as an additional treatment option and to assess long-term effects of BET. Beside the standard procedure, children (4 to 10 years of age), with equal pathology on both ears, will be assigned for BET on side.

DETAILED DESCRIPTION:
Introduction:

Otitis media with effusion (OME, "glue ear") is very common in children and characterized by fluid in the middle ear without signs or symptoms of acute ear infection. Fluid in the middle ear causes conducting hearing loss. OME has a large impact on health care costs and recurrent or persistent OME can effect the proper development of children. Frequently OME resolves itself, therefore guidelines strongly recommend watchful waiting for 3 months after which treatment options are tympanostomy tubes and/or adenoidectomy. However OME often reoccurs after these procedures. Furthermore there are various short and longterm side-effects of tympanostomy tubes.In Balloon Eustachian Tuboplasty (BET) a ballon catheter is used to dilate the cartilage part of the eustachian tube and is inserted through the nose to reach the opening of the tube, located in the nasopharynx. BET has recently been applied in children for therapy-resistant recurrent OME and inflammatory ear diseases with promising results. Risk and complications rates are very low.

Methods:

Goal of this study will be the evaluation of Balloon Eustachian Tuboplasty (BET) in children as a primary treatment of OME. Children between the ages of 4 and 10 years with OME and tympanometry type B on both ears, will prospectively be recruited and assigned for adenoidectomy and myringotomy. Parents then will be asked for participation in this trial and fully informed about purpose, technique and possible side effects. If consent is given, adenoidectomy, in case of large adenoids, and myringotomy will be performed on both sides. If necessary (very thick fluid) tympanostomy tubes are placed. One Eustachian tube of each patient is randomly assigned for BET.

ELIGIBILITY:
Inclusion Criteria:

* OME on both sides measured by flat tympanometry

Exclusion Criteria:

* Patients with cleft lip and/or palate and other severe craniofacial abnormalities

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-12-14 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Tympanometry-Change (Middle ear effusion/eardrum mobility assessed with Tympanometry) | up to 3 months preoperatively and change to 3, 6 and 9 months postoperatively;
  Tympanometry, an objective test of middle-ear function, uses variations of air pressure in the ear canal to assess for middle ear effusion / eardrum mobility.

SECONDARY OUTCOMES:
Otoscopy score | up to 3 months preoperatively and change to 3, 6 and 9 months postoperatively;
  0= no effusion (Valsalva +/-, not feasible)
  1. retracted eardrum
  2. Fluid or bubbles through eardrum visible
  3. complete fluid blockage of middle ear

OTHER OUTCOMES:
symptom-based side depended questionnaire | preoperatively and 9 months postoperatively
  subjective scale side depended (zero to ten points - low to high disturbance by symptom). Symptoms asked for e.g. ear-fullness, pressure, pain, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical university of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeld RM, Shin JJ, Schwartz SR, Coggins R, Gagnon L, Hackell JM, Hoelting D, Hunter LL, Kummer AW, Payne SC, Poe DS, Veling M, Vila PM, Walsh SA, Corrigan MD. Clinical Practice Guideline: Otitis Media with Effusion Executive Summary (Update). Otolaryngol Head Neck Surg. 2016 Feb;154(2):201-14. doi: 10.1177/0194599815624407. PMID 26833645
- [Background] Maier S, Tisch M, Maier H. [Balloon dilation of the Eustachian tube in pediatric chronic obstructive Eustachian tube dysfunction patients]. HNO. 2015 Oct;63(10):686-8, 690-4, 696-7. doi: 10.1007/s00106-015-0050-5. German. PMID 26311130
- [Background] Tisch M, Maier S, Hecht P, Maier H. [Bilateral Eustachian tube dilation in infants: an alternative treatment for persistent middle ear functional dysfunction]. HNO. 2013 Jun;61(6):492-3. doi: 10.1007/s00106-013-2713-4. German. PMID 23712367
- [Background] Popova D, Varbanova S, Popov TM. Comparison between myringotomy and tympanostomy tubes in combination with adenoidectomy in 3-7-year-old children with otitis media with effusion. Int J Pediatr Otorhinolaryngol. 2010 Jul;74(7):777-80. doi: 10.1016/j.ijporl.2010.03.054. PMID 20399511
- [Background] Jenckel F, Kappo N, Gliese A, Loewenthal M, Lorincz BB, Knecht R, Dalchow CV. Endonasal dilatation of the Eustachian tube (EET) in children: feasibility and the role of tubomanometry (Esteve) in outcomes measurement. Eur Arch Otorhinolaryngol. 2015 Dec;272(12):3677-83. doi: 10.1007/s00405-014-3443-2. Epub 2014 Dec 19. PMID 25524643
- [Background] Van Roeyen S, Van de Heyning P, Van Rompaey V. Delayed-Start Study Design for Balloon Dilation of the Eustachian Tube: Alternative for a Randomized Controlled Trial. Front Surg. 2017 Feb 20;4:10. doi: 10.3389/fsurg.2017.00010. eCollection 2017. No abstract available. PMID 28265561
- [Background] Poe D, Anand V, Dean M, Roberts WH, Stolovitzky JP, Hoffmann K, Nachlas NE, Light JP, Widick MH, Sugrue JP, Elliott CL, Rosenberg SI, Guillory P, Brown N, Syms CA 3rd, Hilton CW, McElveen JT Jr, Singh A, Weiss RL Jr, Arriaga MA, Leopold JP. Balloon dilation of the eustachian tube for dilatory dysfunction: A randomized controlled trial. Laryngoscope. 2018 May;128(5):1200-1206. doi: 10.1002/lary.26827. Epub 2017 Sep 20. PMID 28940574